CLINICAL TRIAL: NCT03034447
Title: Obstructive Sleep Apnea in Asthmatic Children: Does the Sex Matter?
Brief Title: Sleep Apnea in Asthmatic Children and Teenagers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Principal Investigator, Gustavo Antonio Moreira, Medical Doctor, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CEP/UNIFESP 1398/2016
Record Dates: First submitted 2017-01-20; First posted 2017-01-27 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Asthma, Bronchial; Bronchial Asthma; Apnea, Sleep; Sleep Apnea, Mixed Central and Obstructive; Sleep Hypopnea (Diagnosis); Obstructive Sleep Apnea; Obstructive Sleep Apnea Syndrome
Keywords: Asthma; Obstructive Sleep Apnea; Children; Teenagers
MeSH Terms: conditions — Asthma; Sleep Apnea Syndromes; Disease; Sleep Apnea, Obstructive | interventions — Surveys and Questionnaires; Respiratory Physiological Phenomena

STUDY DESIGN:
Intervention Model Description: Sleep study and spirometric evaluation of children with asthma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Asthma (Other): Children and teenagers with persistent asthma will perform questionnaires, lung function test, and home sleep study
  Interventions: Other: Questionnaire; Other: Lung Function Test; Other: Home Sleep Study

INTERVENTIONS:
Other: Questionnaire — Children and parents are going to inform data regarding socioeconomical status, asthma and rhinitis diagnosis, asthma and rhinitis control, medications, sleep complaints, and sleep habits
Other: Lung Function Test — Children are going to blow in a machine that measures how the lung is working
  Other Names: Spirometry
Other: Home Sleep Study — Children are going to sleep at home with a device that tells if they stop breathing during sleep
  Other Names: Polysomnography

SUMMARY:
Asthma and sleep apnea are both respiratory diseases and one can worsen the other. Those who suffer from asthma have a higher risk of sleep apnea and sleep apnea can make the asthma more difficult to control.

As girls usually have a more severe asthma than boys, the investigators believe that girls have a higher risk of sleep apnea.

To test if asthmatic girls have more sleep apnea than boys, the investigators are going to ask them questions regarding asthma and sleep symptoms (such as snore) and the investigators are going test the lung function and how many times they stop breathing during the sleep. The sleep test is going to be performed in children's home.

In children, having sleep apnea can make the asthmatic stay in the hospital 30% more when they have an asthma attack. We also are going to look if sleep apnea increases the number of hospitalizations and asthma attacks in the past 12 months.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) and asthma are both inflammatory airway diseases. A systematic review regarding sleep-disordered breathing (SDB) in asthmatic children analyzed 17 studies but only two of them had objective OSA measurement. In total, 45,115 children were included, 53% boys, mean age 8.6 ± 2.5 years. SDB was present in 23.8% of asthmatic children and in 16.7% of non-asthmatic (p < 0.001, OR 1.9, 95%CI 1.7-2.2).

An American study found that OSA in asthmatic children increases hospital length of stay (OR 2.3; 95% CI = 1.8 - 2.9). Brazilian database of the year 2015 showed that, among children 5-19 years, asthma was the 5th cause of hospitalization: a total of 2.4% of the hospitalization in this age group, after birth and its complication (31%), limb fractures (5.7%), pneumonia (3.8%), and appendicitis (3.2%).

The relationship among asthma severity (mild, moderate, and severe) and OSA has been described previously, but not in every study. Poor asthma control has also been linked to a higher OSA risk in adults and children.

OSA and asthma share many risk factors: rhinitis, increased collapsibility of the upper airway, local and systemic inflammation, gastroesophageal reflux, and obesity.

A higher risk of SDB in asthmatic girls has recently been described (OR 2.55 for girls and 0.70 for boys). Among non-asthmatic children OSA is usually equal among boys and girls until adolescence. A possible explanation is asthma severity in children: younger boys are more severe but after puberty, girls are.

Since OSA and asthma are linked diseases and that little is known about them in the pediatric field, specially differences related to sex, the investigators hypothesize that: 1) asthmatic girls have a higher OSA risk; 2) OSA will be higher in asthmatic children compared to the pediatric literature; 3) asthma severity, asthma control, and rhinitis will be related to a higher OSA risk. The investigators also aim to analyze factors associated with a higher risk of hospitalizations and asthma attacks.

ELIGIBILITY:
Inclusion Criteria:

* Persistent asthma

Exclusion Criteria:

* Craniofacial malformation
* Thoracic malformation
* Genetic syndromes
* Bronchopulmonary dysplasia
* Bronchiolitis obliterans
* Neuromuscular diseases
* Sickle cell anemia
* Cystic fibrosis

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-12; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Sleep Apnea Syndrome | 1 night
  Apneas and hypopneas during sleep

SECONDARY OUTCOMES:
Asthma Control | 4 weeks
  Asthma Control based on Global Initiative for Asthma (GINA) questions
ER visits | 1 year
  How many times went to hospital the previous year
Lung function | 1 day
  Currently lung function

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo A Moreira, MD, Study Chair — Federal University of São Paulo
Locations (1):
- Federal University of São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Malakasioti G, Gourgoulianis K, Chrousos G, Kaditis A. Interactions of obstructive sleep-disordered breathing with recurrent wheezing or asthma and their effects on sleep quality. Pediatr Pulmonol. 2011 Nov;46(11):1047-54. doi: 10.1002/ppul.21497. Epub 2011 Aug 1. PMID 21809473
- [Background] Kheirandish-Gozal L, Dayyat EA, Eid NS, Morton RL, Gozal D. Obstructive sleep apnea in poorly controlled asthmatic children: effect of adenotonsillectomy. Pediatr Pulmonol. 2011 Sep;46(9):913-8. doi: 10.1002/ppul.21451. Epub 2011 Apr 4. PMID 21465680
- [Background] Alonso-Alvarez ML, Teran-Santos J, Ordax Carbajo E, Cordero-Guevara JA, Navazo-Eguia AI, Kheirandish-Gozal L, Gozal D. Reliability of home respiratory polygraphy for the diagnosis of sleep apnea in children. Chest. 2015 Apr;147(4):1020-1028. doi: 10.1378/chest.14-1959. PMID 25539419
- [Background] Shanley LA, Lin H, Flores G. Factors associated with length of stay for pediatric asthma hospitalizations. J Asthma. 2015 Jun;52(5):471-7. doi: 10.3109/02770903.2014.984843. Epub 2014 Nov 21. PMID 25375904
- [Background] Goldstein NA, Aronin C, Kantrowitz B, Hershcopf R, Fishkin S, Lee H, Weaver DE, Yip C, Liaw C, Saadia TA, Abramowitz J, Weedon J. The prevalence of sleep-disordered breathing in children with asthma and its behavioral effects. Pediatr Pulmonol. 2015 Nov;50(11):1128-36. doi: 10.1002/ppul.23120. Epub 2014 Dec 2. PMID 25461921